CLINICAL TRIAL: NCT06532006
Title: A Randomized, Double-blinded, Multicenter, Phase Ⅲ Clinical Study of HLX22 (Recombinant Humanized Anti-HER2 Monoclonal Antibody Injection) in Combination With Trastuzumab and Chemotherapy (XELOX) Versus Trastuzumab and Chemotherapy (XELOX) With or Without Pembrolizumab for the First Line Treatment of Locally Advanced or Metastatic Gastroesophageal Junction and Gastric Cancer
Brief Title: A Phase Ⅲ Clinical Study of HLX22 in Combination With Trastuzumab and Chemotherapy for the Treatment of Gastroesophageal Junction and Gastric Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Collaborators: Henlius USA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX22-GC-301
Record Dates: First submitted 2024-07-25; First posted 2024-08-01 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-01

CONDITIONS: Gastroesophageal-junction Cancer; Monoclonal Antibody; Gastric Cancer; HER2-positive Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — pembrolizumab; Trastuzumab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group: HLX22 (15 mg/kg) + trastuzumab + chemotherapy (XELOX) ± placebo (for pembrolizumab), Q3W
  Subjects in the experimental group may use one of the treatments below:
  HLX22 (15 mg/kg) + trastuzumab + chemotherapy (XELOX) or HLX22 (15 mg/kg) + trastuzumab + chemotherapy (XELOX) + placebo (for pembrolizumab)
  Interventions: Drug: HLX22; Drug: Trastuzumab; Drug: Oxaliplatin; Drug: Capecitabine
- Control group (Active Comparator): Control group: Placebo (for HLX22) + trastuzumab + chemotherapy (XELOX) ± pembrolizumab, Q3W
  Subjects in the control group may use one of the treatments below:
  Placebo (for HLX22) + trastuzumab + chemotherapy (XELOX) or Placebo (for HLX22) + trastuzumab + chemotherapy (XELOX) + pembrolizumab
  Interventions: Drug: Pembrolizumab; Drug: Trastuzumab; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: HLX22 — HLX22 15mg/kg Q3w
  Arms: Experimental group
Drug: Pembrolizumab — Pembrolizumab 200mg q3w
  Arms: Control group
Drug: Trastuzumab — Trastuzumab 8 mg/kg loading dose and then 6 mg/kg maintenance thereafter ,Q3W
Drug: Oxaliplatin — Oxaliplatin 130 mg/m2 ,Q3W
Drug: Capecitabine — Capecitabine 1000 mg/m2 bid on Days 1-14 ,Q3W

SUMMARY:
This is a double-blind, randomized, multiregion, comparative phase Ⅲ clinical study designed to evaluate the efficacy and safety of HLX22 in combination with trastuzumab and chemotherapy as first-line treatment in patients with HER2-positive locally advanced/metastatic adenocarcinoma of the gastric and/or gastroesophageal junction (G/GEJ).Eligible subjects will be randomized to the two groups based on a 1:1 ratio. Enrolled subjects shall be treated with the study drug until the loss of clinical benefit, death, intolerable toxicity, withdrawal of informed consent, or other reasons specified by the protocol (whichever occurs first).

DETAILED DESCRIPTION:
In experimental group: HLX22 (15 mg/kg) + trastuzumab + chemotherapy (XELOX) ± placebo (for pembrolizumab), once every 3 weeks (Q3W).

In control group: Placebo (for HLX22) + trastuzumab + chemotherapy (XELOX) ± pembrolizumab, Q3W.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female who are at least 18 years of age on the day of signing the informed consent.
2. With histologically or cytologically confirmed diagnosis of previously untreated, locally advanced unresectable or metastatic HER2-positive gastric or gastroesophageal junction adenocarcinoma.
3. Had measurable disease as assessed by IRRC according to the RECIST v1.1, the target lesion must not be a bone metastatic lesion only.
4. HER2-positive tumor defined as either IHC 3+ or IHC 2+ in combination with ISH+ or FISH, as assessed by a central laboratory on a primary or metastatic tumor.
5. ECOG PS within 7 days before randomization: 0-1.
6. Expected survival ≥ 6 months.
7. Had adequate organ function

Exclusion Criteria:

1. Patients with other malignant tumors within 2 years before the randomization.
2. Evidence of disease progression within 6 months (before randomization) after completion of prior neoadjuvant or adjuvant chemotherapy (or both) or radiotherapy for gastric adenocarcinoma or gastroesophageal junction adenocarcinoma.
3. Previous treatment with any HER2-target therapy.
4. Active gastrointestinal bleeding
5. Presence of central nervous system (CNS) metastases.
6. Left ventricular ejection fraction (LVEF) < 55%.
7. Subjects who had known history of severe allergy to any monoclonal antibody or any component of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS)per RECIST 1.1 assessed by IRRC(Independent Radiology Review Committee) | Up to 5 years
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 or death due to any cause, whichever occurs first. PFS will be determined for each treatment arm
Overall Survival （OS） | Up to 5 years
  OS is defined as the time from randomization to death due to any cause. OS will be determined for each treatment arm.

SECONDARY OUTCOMES:
PFS per RECIST 1.1 assessed by investigator | Up to 5 years
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 or death due to any cause, whichever occurs first. PFS will be determined for each treatment arm
Objective Response Rate (ORR) assessed by IRRC and investigator per RECIST v1.1 | Up to 5 years
  ORR is defined as the percentage of participants who have a Complete Response ([CR], disappearance of all evidence of disease) or Partial Response ([PR], regression of measurable disease and no new sites) per RECIST 1.1. ORR will be determined for each treatment arm.
Adverse events (AE) | Up to 5 years
  An AE is any untoward medical occurrence in a participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. The number of participants who experience an AE will be reported for each treatment arm.

CONTACTS AND LOCATIONS:
Locations (88):
- United States (26):
  - Los Angeles Cancer Network, Anaheim, California
  - OPN - Oncology Physician Network (Los Alamitos), Los Alamitos, California
  - Banner MD Anderson Cancer Center, Greeley, Colorado
  - Advanced Research LLC, Deerfield Beach, Florida
  - Florida Cancer Specialist - South, Fort Myers, Florida
  - BRCR Medical Center, Plantation, Florida
  - Napa Research, Pompano Beach, Florida
  - Florida Cancer Specialist - North, St. Petersburg, Florida
  - Florida Cancer Specialist - East, West Palm Beach, Florida
  - Northwestern University, Chicago, Illinois
  - Mission Cancer + Blood (Exigent Network), Des Moines, Iowa
  - Holden Comprehensive Cancer Center - University of Iowa, Iowa City, Iowa
  - Washington University School of Medicine St. Louis, St Louis, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Centers Nevada, Las Vegas, Nevada
  - Cleveland Clinic, Cleveland, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Guthrie Medical Group, PC and Robert Packer Hospital (Guthrie Cancer Center - Sayre), Sayre, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology - West (SCRI), Abilene, Texas
  - Texas Oncology Central South (SCRI), Austin, Texas
  - The University of Texas MD Anderson cancer Center, Houston, Texas
  - Texas Oncology - Gulf Coast (SCRI), Webster, Texas
  - American Oncology Network Vista Oncology Division, Olympia, Washington
  - Northwest Medical Specialties, Tacoma, Washington
  - West Virginia University Cancer Institute, Morgantown, West Virginia
- Australia (7):
  - St. Vincent Hospital Melbourne, Fitzroy, Melbourne
  - Peninsula Health-Frankston hospital, Frankston, Melbourne
  - University of the Sunshine Coast Clinical Trials, Sunshine Coast Haematology and Oncology Clinic, Sunshine Coast, Queensland
  - GenesisCare Research, Campbelltown, Sydney
  - Central Coast Local Health District (Gosford and Wyong Hospital), Gosford, Sydney
  - Macquarie University, North Ryde, Sydney
  - Concord Repatriation General Hospital, Concord
- Chile (2):
  - Centro de Oncologia de Precision, Santiago, Santiago Metropolitan
  - Instituto del Cancer RedSalud Vitacura, Santiago, Santiago Metropolitan
- China (43):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Affiliated Hospital of Youjiang Medical University for Nationalities, Baise City
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu
  - The First Hospital of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi
  - Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, Chengdu
  - West China Hospital of Sichuan University, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Fujian Cancer Hospital, Fuzhou
  - Zhongshan City People's Hospital, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - Sir Run Run Shaw Hospital (SRRSH), affiliated with the Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital, Zhejiang University School of Medic, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - The Second Hospital of Anhui Medical University, Hefei
  - Cancer Hospital of Shandong First Medical University, Jinan
  - Gansu Provincial Cancer Hospital, Lanzhou
  - Gansu Provincial Hospital, Lanzhou
  - The First Hospital Of Lanzhou University, Lanzhou
  - Liuzhou Workers' Hospital, Liuchow
  - The First Affiliated Hospital of Henan University of Science, Luoyang
  - Mianyang Central Hospital, Mianyang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Renji Hospital,Shanghai Jiao Tong University School of Medicine, Shanghai
  - The Central Hospital of Shaoyang, Shaoyang
  - Liaoning Medical University Cancer Institute & Hospital, Shenyang
  - Shanxi Cancer Hospital, Taiyuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Cancer Hospital Affiliated to Xinjiang Medical University, Ürümqi
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Qinghai University Affiliated Hospital, Xining
  - Xuzhou Central Hospital, Xuzhou
  - Yichang Central People's Hospital, Yichang
  - General Hospital of Ningxia Medical University, Yinchuan
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- Georgia (5):
  - LLC Todua Clinic, Tbilisi
  - Ltd "New Hospitals", Tbilisi
  - Tbilisi State Medical University and Ingorovka High Medical Technology University Clinic Ltd, Tbilisi
  - JSV VIAN- Caraps Medline, Tbilisi
  - Evex Hospitals - Caucasus Medical Center, Tbilisi
- Japan (5):
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Ishikawa Prefectural Central Hospital, Kanazawa
  - Osaki Citizen Hospital, Osaki-shi
  - Saitama Cancer Center, Saitama
  - Keiyukai Sapporo Hospital, Sapporo

IPD SHARING:
Plan to Share IPD: No